CLINICAL TRIAL: NCT00340210
Title: Extended Follow-up of Columbia, MO Serum Bank Participants
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999999002; OH99-C-N002
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer; Endometrial Cancer; Ovarian Cancer
Keywords: Biomarkers; Breast Cancer; Etiology; Hormones; Prospective Study
MeSH Terms: conditions — Breast Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Serum Bank Participants: The Columbia MO Serum Bank recruited 6915 women living in and around Columbia MO between 1977-1987 who were cancer-free except for non-melanoma skin cancer and at least 18 years of age.

SUMMARY:
The Columbia, MO Serum Bank initially was established in 1977 as part of the National Cancer Institute's (NCI) Biological Markers Project to identify serum markers for breast cancer. Participants were volunteers identified through the Breast Cancer Detection Demonstration Project (BCDDP) at the University of Missouri Hospital and Ellis Fischel Cancer Center in Columbia, MO. A total of 6,915 women without a prior history of cancer, other than non-melanoma skin cancer, donated blood to the bank on one or more occasions between 1977 and 1987.

At the time of each blood collection, interview information was obtained including age, height, weight, reproductive and menstrual histories, family history of breast cancer, medical conditions, and drug use, including oral contraceptives and menopausal hormone therapy. Date of last menstrual period was captured for women who were premenopausal at the time of each blood collection. Approximately 30% of the women donated multiple samples over the first 10 years of the study, (including 20% with 3 or more samples), with collections occurring on average one year apart. At each collection, serum was aliquoted into up to ten, 1 ml vials and stored at -70 (Infinite)C at the NCI Repository. All women gave informed consent before donating to the serum bank.

The initial follow-up continued for up to 12 years through 1989, with 244 cancers identified. Of the 6915 original participants, 79% were last seen in 1983 or earlier, yielding a median follow-up time of 4 years. A questionnaire was mailed to all participants annually to ascertain information on interim breast biopsies and cancer diagnoses. Women who indicated that they had a breast biopsy or breast cancer were sent a consent form for permission to obtain medical records including pathology reports. For cancers at sites other than the breast, medical records and pathology reports were not requested, although date of diagnosis and site were ascertained.

Between 1999 and 2002, an extended follow-up of Columbia, MO Serum Bank participants was conducted. Of the 6915 original participants, 6,720 women had blood remaining and were included in this phase of the study. Of these, 6,154 (91.6%) were located; 566 (8%) were not locatable, 109 (2%) refused to participate, and 40 (<1%) were too ill to participate. 1,694 women (25%) were deceased. This last follow-up identified an additional 1123 cancers. This cohort has serum samples from a cohort of 6720 pre- and postmenopausal women followed up to 20 years for cancer diagnoses and is a unique resource for molecular epidemiologic studies exploring serum markers associated with cancer risk.

DETAILED DESCRIPTION:
The Columbia, MO Serum Bank initially was established in 1977 as part of the National Cancer Institute's (NCI) Biological Markers Project to identify serum markers for breast cancer. Participants were volunteers identified through the Breast Cancer Detection Demonstration Project (BCDDP) at the University of Missouri Hospital and Ellis Fischel Cancer Center in Columbia, MO. A total of 6,915 women without a prior history of cancer, other than non-melanoma skin cancer, donated blood to the bank on one or more occasions between 1977 and 1987.

At the time of each blood collection, interview information was obtained including age, height, weight, reproductive and menstrual histories, family history of breast cancer, medical conditions, and drug use, including oral contraceptives and menopausal hormone therapy. Date of last menstrual period was captured for women who were premenopausal at the time of each blood collection. Approximately 30% of the women donated multiple samples over the first 10 years of the study, (including 20% with 3 or more samples), with collections occurring on average one year apart. At each collection, serum was aliquoted into up to ten, 1 ml vials and stored at -70 (Infinite)C at the NCI Repository. All women gave informed consent before donating to the serum bank.

The initial follow-up continued for up to 12 years through 1989, with 244 cancers identified. Of the 6915 original participants, 79% were last seen in 1983 or earlier, yielding a median follow-up time of 4 years. A questionnaire was mailed to all participants annually to ascertain information on interim breast biopsies and cancer diagnoses. Women who indicated that they had a breast biopsy or breast cancer were sent a consent form for permission to obtain medical records including pathology reports. For cancers at sites other than the breast, medical records and pathology reports were not requested, although date of diagnosis and site were ascertained.

Between 1999 and 2002, an extended follow-up of Columbia, MO Serum Bank participants was conducted. Of the 6915 original participants, 6,720 women had blood remaining and were included in this phase of the study. Of these, 6,154 (91.6%) were located; 566 (8%) were not locatable, 109 (2%) refused to participate, and 40 (<1%) were too ill to participate. 1,694 women (25%) were deceased. This last follow-up identified an additional 1123 cancers. This cohort has serum samples from a cohort of 6720 pre- and postmenopausal women followed up to 20 years for cancer diagnoses and is a unique resource for molecular epidemiologic studies exploring serum markers associated with cancer risk.

ELIGIBILITY:
* Not listed.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Columbia MO Serum Bank recruited 6915 women living in and around Columbia MO between 1977- 1987 who were cancer-free except for non-melanoma skin cancer and at least 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 6720 (Actual)
Dates: Start 1999-01-14 (Actual); Primary Completion 2014-06-24 (Actual); Study Completion 2014-09-02 (Actual)

PRIMARY OUTCOMES:
Primary Cancer diagnosis | time of diagnosis
  Primary Cancer diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Benson, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dorgan JF, Longcope C, Stephenson HE Jr, Falk RT, Miller R, Franz C, Kahle L, Campbell WS, Tangrea JA, Schatzkin A. Relation of prediagnostic serum estrogen and androgen levels to breast cancer risk. Cancer Epidemiol Biomarkers Prev. 1996 Jul;5(7):533-9. PMID 8827358
- [Background] Dorgan JF, Stanczyk FZ, Longcope C, Stephenson HE Jr, Chang L, Miller R, Franz C, Falk RT, Kahle L. Relationship of serum dehydroepiandrosterone (DHEA), DHEA sulfate, and 5-androstene-3 beta, 17 beta-diol to risk of breast cancer in postmenopausal women. Cancer Epidemiol Biomarkers Prev. 1997 Mar;6(3):177-81. PMID 9138660
- [Background] Falk RT, Dorgan JF, Kahle L, Potischman N, Longcope C. Assay reproducibility of hormone measurements in postmenopausal women. Cancer Epidemiol Biomarkers Prev. 1997 Jun;6(6):429-32. PMID 9184776